CLINICAL TRIAL: NCT01516099
Title: Pilot Study: A Structural Approach to Implement the Role of 'Physical Activity Counselors' in Sports and Exercise Promotion in Flanders
Brief Title: A Structural Approach to Implement the Role of 'Physical Activity Counselors' in Sports and Exercise Promotion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgian Government (Other Government)
Responsible Party: Principal Investigator, Christophe Delecluse, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S53801
Record Dates: First submitted 2012-01-12; First posted 2012-01-24 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Sedentary Lifestyle
Keywords: Physical activity counselor; Active and healthy lifestyle; General Practitioner; Social-cultural Organization
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — General Practitioners

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Practitioners (Experimental): The general practitioner can refer his patients to a physical activity counselor for an individual coaching. The investigators aim for a brief coaching period of 10 weeks with the objective that the people continue their active lifestyle afterwards.
  Interventions: Other: General Practitioners
- Social-cultural organizations (Experimental): In the social-cultural organization, members can sign in for group sessions led by the physical activity counselor. The investigators aim for a brief coaching period of 10 weeks with the objective that the people continue their active lifestyle afterwards.
  Interventions: Other: Social-cultural organizations

INTERVENTIONS:
Other: General Practitioners — The general practitioner can refer his patients to a physical activity counselor for an individual coaching (intake session with development of program and pretesting, follow up by e-mail or phone (max 4x), personal contact moments (max 3x) and exit session with evaluation and posttesting).
  Arms: General Practitioners
Other: Social-cultural organizations — In the social-cultural organization, members can sign in for group sessions led by the physical activity counselor (intake session with development of program and pretesting, follow up by email or letters (max 4x), personal contact moments (max 4x) and exit session with evaluation and posttesting).
  Arms: Social-cultural organizations

SUMMARY:
The primary aim of this study is to investigate how a physical activity counselor can offer an added value in the sports and exercise promotion in Flanders. The investigators will explore if the physical activity counselor, in collaboration with the setting of general practitioners and social-cultural associations, can refer sedentary people and persons who are active in a non-organized context, into systematic participation in sports and/or exercise. Additionally, the investigators want to determine if the physical activity counselor will succeed in referring the target population to the local supervised and structured sports and exercise activities.

DETAILED DESCRIPTION:
Being regularly physically active is a basic component of a healthy lifestyle. However, a large amount of the Flemish population does not reach the prescribed guidelines and cannot enjoy the health benefits related to an active lifestyle. One part of the population is physically active but makes no use of the existing, structured and supervised exercise and sports programs. Therefore the chance on lifetime participation in sports and exercise is quite low in this group. Another group consists of sedentary people that does not participate in any exercise or sports activity at all.

A physical activity counselor can possibly deliver a crucial service for the above mentioned groups. He/she can design an individualized sports- or exercise approach and program. In the short term, the physical activity counselor can guide the participant into his first success experiences regarding exercise and sports. In the long term, the chance of remaining physically active will increase by improving the understanding and the self-confidence of these participants.

However it is questioned how the physical activity counselor can reach these target groups in an efficient way, as the traditional sports and exercise promotion seems to have no impact on these persons. A first alternative may be the setting of the general practitioners. The general practitioner is, as a care provider in primary health care, in a good position to refer sedentary people or those who are active in a non-organized context to a physical activity counselor for 'minimal' coaching. A second alternative can be the setting of the social-cultural associations (e.g. seniors association, women association, neighborhood actions, …). The social context and the local networks in these associations facilitate the proper forms of motivation to exercise with other people and to adapt to a healthy lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-75 years of age
* Able to walk

Exclusion Criteria:

* Severe cardial disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in health-related anthropometric measures | baseline, 10 weeks, 6 months
  Length, Weight, Abdominal circumference
Change in objective measure of degree of physical activity | Baseline, 10 weeks, 6 months
  Sensewear: little accelerometer that will be carried on the upper arm during several days and consequently registrates the amount of physical activity during this period.
Change in mental well-being | Baseline, 10 weeks, 6 months
  Standardized questionnaire
Change in motivation to be physically active | Baseline, 10 weeks, 6 months
  Standardized questionnaire
Change in participation in local structured sports and exercise | Baseline, 10 weeks, 6 months
  Standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Delecluse, PhD, Dr, Principal Investigator — Faculty of Kinesiology and Rehabilitation Sciences
Locations (1):
- Katholieke Universiteit Leuven - Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Vlaams Brabant, Belgium